CLINICAL TRIAL: NCT04485234
Title: Inclusive Invasive Physiological Assessment in Angina Syndromes Registry (ILIAS Registry)
Brief Title: Inclusive Invasive Physiological Assessment in Angina Syndromes Registry
Acronym: ILIAS Registry
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Tergooi Hospital (Other); Amphia Hospital (Other); Seoul National University Hospital (Other); Samsung Medical Center (Other); Inje University (Other); Keimyung University Dongsan Medical Center (Other); Ulsan University Hospital (Other); Tsuchiura Kyodo General Hospital (Other); Hospital San Carlos, Madrid (Other); Aarhus University Hospital (Other); Catholic University of the Sacred Heart (Other); University of Cincinnati (Other); Gifu Heart Center (Other); Toda Central General Hospital (Unknown)
Responsible Party: Principal Investigator, Tim van de Hoef, M.D., Ph.D., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: ILIAS Registry
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease; Microvascular Coronary Artery Disease
Keywords: Coronary flow reserve; Fractional flow reserve; Microvascular resistance; Thermodilution; Doppler flow velocity
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: All lesions undergo assessment with coronary pressure sensor and either Doppler velocity or coronary thermodilution
  Interventions: Diagnostic Test: Resting distal coronary to aortic pressure ratio, Fractional flow reserve, Coronary Flow Reserve, Microvascular resistance

INTERVENTIONS:
Diagnostic Test: Resting distal coronary to aortic pressure ratio, Fractional flow reserve, Coronary Flow Reserve, Microvascular resistance — Calculation of the resting mean distal coronary to aortic pressure ratio (resting Pd/Pa), fractional flow reserve (Pd/Pa at hyperemia), Coronary flow reserve (peak flow/resting flow), microvascular resistance (Pd/flow).

SUMMARY:
This study evaluates the prognostic value and potential therapeutic impact of combined pressure and flow measurements in the evaluation of epicardial coronary stenosis and microvascular function.

DETAILED DESCRIPTION:
ILIAS registry is a global effort to gather lesion-level data on the diagnostic and prognostic value of combined coronary pressure and flow measurements in clinical practice. Data is gathered from 7 nations (The Netherlands, Korea, Japan, Spain, Italy, Denmark, USA), using either coronary Doppler velocity measurements or coronary thermodilution measurements to obtain invasive coronary flow assessment. Patient treatment was governed by the local clinical practice guidelines at the time of the invasive procedure, but was at the operator's discretion. A standardized data collection sheet was used and all study adopted standardized definition of patient's baseline characteristics, clinical outcomes, and physiologic data. In case of acute coronary syndrome (unstable angina, non-ST-segment elevation myocardial infarction, and ST-segment elevation myocardial infarction), only non-culprit vessel evaluation was used.

ELIGIBILITY:
Inclusion Criteria:

* underwent combined measurements of coronary pressure and flow for at least 1native coronary artery

Exclusion Criteria:

* hemodynamic instability
* culprit vessel of acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing clinically indicated invasive coronary angiography and with an indication for invasive physiological evaluation of at least 1 native coronary artery.
Sampling Method: Non-Probability Sample
Enrollment: 2322 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 10 years
  Cumulative incidence of a composite of any death, any myocardial infarction, or any ischemia-driven revascularization

SECONDARY OUTCOMES:
Target vessel failure | 10 years
  Cumulative incidence of a composite of cardiac death, target-vessel related myocardial infarction, or target-vessel revascularization
Individual components of MACE and TVF | 10 years
  Cumulative incidence of the individual components of MACE and TVF

CONTACTS AND LOCATIONS:
Locations (12):
- Cincinnati University Medical Center, Cincinnati, Ohio, United States
- Aarhus University Hospital, Aarhus, Denmark
- Catholic University of the Sacred Heart, Roma, Italy
- Japan (3):
  - Gifu Heart Center, Gifu
  - Toda Central General Hospital, Toda
  - Tsuchiura Kyodo General Hospital, Tsuchiura
- Netherlands (3):
  - Amsterdam UMC - location AMC, Amsterdam
  - Tergooi, Blaricum
  - Amphia Hospital, Breda
- South Korea (2):
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
Anonymized patient level data will be made available by the corresponding author for reasonable requests. Consent was not obtained for data sharing but the presented data are fully anonymized and risk of identification is negligible.

REFERENCES:
- [Derived] Boerhout CKM, Echavarria-Pinto M, de Waard GA, Lee JM, Mejia-Renteria H, Hun Lee S, Jung JH, Hoshino M, Matsuo H, Madera-Cambero M, Eftekhari A, Effat MA, Murai T, Marques K, Doh JH, Christiansen EH, Banerjee R, Nam CW, Niccoli G, Nakayama M, Tanaka N, Shin ES, Beijk MAM, van Royen N, Knaapen P, Escaned J, Kakuta T, Koo BK, Piek JJ, van de Hoef TP, Meuwissen M. Impact of hyperaemic stenosis resistance on long-term outcomes of stable angina in the ILIAS Registry. EuroIntervention. 2024 Jun 3;20(11):e699-e706. doi: 10.4244/EIJ-D-23-00713. PMID 38840578
- [Derived] Vink CEM, Woudstra J, Lee JM, Boerhout CKM, Cook CM, Hoshino M, Mejia-Renteria H, Lee SH, Jung JH, Echavarria-Pinto M, Meuwissen M, Matsuo H, Madera-Cambero M, Eftekhari A, Effat MA, Murai T, Marques K, Beijk MAM, Doh JH, Piek JJ, van de Hoef TP, Christiansen EH, Banerjee R, Nam CW, Niccoli G, Nakayama M, Tanaka N, Shin ES, van Royen N, Chamuleau SAJ, Knaapen P, Escaned J, Kakuta T, Koo BK, Appelman Y, de Waard GA. Sex differences in prevalence and outcomes of the different endotypes of chronic coronary syndrome in symptomatic patients undergoing invasive coronary angiography: Insights from the global ILIAS invasive coronary physiology registry. Atherosclerosis. 2023 Nov;384:117167. doi: 10.1016/j.atherosclerosis.2023.06.073. Epub 2023 Jul 8. PMID 37558604
- [Derived] Hoshino M, van de Hoef TP, Lee JM, Hamaya R, Kanaji Y, Boerhout CKM, de Waard GA, Jung JH, Lee SH, Mejia-Renteria H, Echavarria-Pinto M, Meuwissen M, Matsuo H, Madera-Cambero M, Eftekhari A, Effat MA, Marques K, Doh JH, Christiansen EH, Banerjee R, Nam CW, Niccoli G, Murai T, Nakayama M, Tanaka N, Shin ES, Sasano T, Appelman Y, Beijk M, Knaapen P, van Royen N, Escaned J, Koo BK, Piek JJ, Kakuta T. Abnormal physiological findings after FFR-based revascularisation deferral are associated with worse prognosis in women. Sci Rep. 2023 Jan 19;13(1):1027. doi: 10.1038/s41598-023-28146-6. PMID 36658168
- [Derived] Boerhout CKM, de Waard GA, Lee JM, Mejia-Renteria H, Lee SH, Jung JH, Hoshino M, Echavarria-Pinto M, Meuwissen M, Matsuo H, Madera-Cambero M, Eftekhari A, Effat MA, Murai T, Marques K, Doh JH, Christiansen EH, Banerjee R, Nam CW, Niccoli G, Nakayama M, Tanaka N, Shin ES, Chamuleau SAJ, van Royen N, Knaapen P, Escaned J, Kakuta T, Koo BK, Piek JJ, van de Hoef TP. Combined use of hyperemic and non-hyperemic pressure ratios for revascularization decision-making: From the ILIAS registry. Int J Cardiol. 2023 Jan 1;370:105-111. doi: 10.1016/j.ijcard.2022.11.015. Epub 2022 Nov 11. PMID 36372287
- [Derived] Joh HS, Shin D, Lee JM, Lee SH, Hong D, Choi KH, Hwang D, Boerhout CKM, de Waard GA, Jung JH, Mejia-Renteria H, Hoshino M, Echavarria-Pinto M, Meuwissen M, Matsuo H, Madera-Cambero M, Eftekhari A, Effat MA, Murai T, Marques K, Doh JH, Christiansen EH, Banerjee R, Kim HK, Nam CW, Niccoli G, Nakayama M, Tanaka N, Shin ES, Chamuleau SAJ, van Royen N, Knaapen P, Koo BK, Kakuta T, Escaned J, Piek JJ, van de Hoef TP; ILIAS Registry Investigators [Link]. Prognostic Impact of Coronary Flow Reserve in Patients With Reduced Left Ventricular Ejection Fraction. J Am Heart Assoc. 2022 Aug 2;11(15):e025841. doi: 10.1161/JAHA.122.025841. Epub 2022 Jul 25. PMID 35876408
- [Derived] Boerhout CKM, de Waard GA, Lee JM, Mejia-Renteria H, Lee SH, Jung JH, Hoshino M, Echavarria-Pinto M, Meuwissen M, Matsuo H, Madera-Cambero M, Eftekhari A, Effat MA, Murai T, Marques K, Appelman Y, Doh JH, Christiansen EH, Banerjee R, Nam CW, Niccoli G, Nakayama M, Tanaka N, Shin ES, Beijk MAM, Knaapen P, Escaned J, Kakuta T, Koo BK, Piek JJ, van de Hoef TP. Prognostic value of structural and functional coronary microvascular dysfunction in patients with non-obstructive coronary artery disease; from the multicentre international ILIAS registry. EuroIntervention. 2022 Oct 21;18(9):719-728. doi: 10.4244/EIJ-D-22-00043. PMID 35694826
- [Derived] van de Hoef TP, Lee JM, Boerhout CKM, de Waard GA, Jung JH, Lee SH, Mejia-Renteria H, Hoshino M, Echavarria-Pinto M, Meuwissen M, Matsuo H, Madera-Cambero M, Eftekhari A, Effat MA, Murai T, Marques K, Doh JH, Christiansen EH, Banerjee R, Nam CW, Niccoli G, Nakayama M, Tanaka N, Shin ES, van Royen N, Chamuleau SAJ, Knaapen P, Escaned J, Kakuta T, Koo BK, Piek JJ. Combined Assessment of FFR and CFR for Decision Making in Coronary Revascularization: From the Multicenter International ILIAS Registry. JACC Cardiovasc Interv. 2022 May 23;15(10):1047-1056. doi: 10.1016/j.jcin.2022.03.016. PMID 35589234
- [Derived] Kim J, Shin D, Lee JM, Lee SH, Hong D, Choi KH, Hwang D, Boerhout CKM, de Waard GA, Jung JH, Mejia-Renteria H, Hoshino M, Echavarria-Pinto M, Meuwissen M, Matsuo H, Madera-Cambero M, Eftekhari A, Effat MA, Murai T, Marques K, Doh JH, Christiansen EH, Banerjee R, Kim HK, Nam CW, Niccoli G, Nakayama M, Tanaka N, Shin ES, Chamuleau SAJ, van Royen N, Knaapen P, Koo BK, Kakuta T, Escaned J, Piek JJ, van de Hoef TP; ILIAS Registry Investigators. Differential Prognostic Value of Revascularization for Coronary Stenosis With Intermediate FFR by Coronary Flow Reserve. JACC Cardiovasc Interv. 2022 May 23;15(10):1033-1043. doi: 10.1016/j.jcin.2022.01.297. Epub 2022 Apr 27. PMID 35490124
- [Derived] Lee SH, Shin D, Lee JM, van de Hoef TP, Hong D, Choi KH, Hwang D, Boerhout CKM, de Waard GA, Jung JH, Mejia-Renteria H, Hoshino M, Echavarria-Pinto M, Meuwissen M, Matsuo H, Madera-Cambero M, Eftekhari A, Effat MA, Murai T, Marques K, Doh JH, Christiansen EH, Banerjee R, Kim HK, Nam CW, Niccoli G, Nakayama M, Tanaka N, Shin ES, Chamuleau SAJ, van Royen N, Knaapen P, Koo BK, Kakuta T, Escaned J, Piek JJ; ILIAS Registry Investigators dagger. Clinical Relevance of Ischemia with Nonobstructive Coronary Arteries According to Coronary Microvascular Dysfunction. J Am Heart Assoc. 2022 May 3;11(9):e025171. doi: 10.1161/JAHA.121.025171. Epub 2022 Apr 27. PMID 35475358